CLINICAL TRIAL: NCT00847366
Title: An Open Label Trial of Perifosine in Patients Currently Being Treated on Perifosine Trials in Solid Tumors or Multiple Myeloma
Brief Title: Open Label Trial of Perifosine in Patients Currently Being Treated on Perifosine Trials in Solid Tumors or Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 534
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-02

CONDITIONS: Non Small Cell Lung Cancer; Solid Tumors; Metastatic Breast Cancer; Sarcomas
Keywords: Perifosine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Sarcoma | interventions — perifosine; Trastuzumab; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Perifosine 201 (Experimental): Perifosine 201: A Phase 1/2 trial of Perifosine in the Treatment of Non-Small Cell Lung Cancer.
  Perifosine dosage:
  Arm A: 50 mg p.o. 3 times daily with meals. Arm B: 150 mg p.o. daily at bedtime. Arm C: 300 mg p.o. 3 times a day (900 mg) once a week.
  Interventions: Drug: Perifosine
- Perifosine 206 (Experimental): Perifosine 206: A Randomized Phase II Trial of Three Doses of Perifosine in Combination with Trastuzumab.
  Arm A: Perifosine 50 mg p.o. daily + 6 mg/kg Trastuzumab on day 1 of a 21-day cycle or 2 mg/kg on days 1, 8 and 15 of a 21 day cycle.
  Arm B: Perifosine 50 mg p.o three times a day + 6 mg/kg Trastuzumab on day 1 of a 21-day cycle or 2 mg/kg on days 1, 8 and 15 of a 21 day cycle.
  Arm C: Perifosine 300 mg three times on one day + 6 mg/kg Trastuzumab on day 1 of a 21-day cycle or 2 mg/kg on days 1, 8 and 15 of a 21 day cycle.
  Interventions: Drug: Perifosine; Drug: Trastuzumab
- Perifosine 207 (Experimental): Perifosine 207: a Phase IIA Trial of Two Schedules of Perifosine Arm A: 50 mg daily with food. Arm B: 50 mg twice daily with food.
  Interventions: Drug: Perifosine
- Perifosine 208 (Experimental): Perifosine 208: A Phase II Trial of Two Schedules of Perifosine in Combination with Endocrine Therapy (Tamoxifen) for Patients with Estrogen Receptor or Progesterone Receptor Positive Metastatic Breast Cancer Dosage: Arm A: 50 mg Perifosine /day p.o. .Endocrine therapy continued at same dose and schedule. Arm B: 900 Perifosine weekly. Endocrine therapy continued at same dose and schedule.
  Interventions: Drug: Perifosine; Drug: Tamoxifen
- Perifosine 209 (Experimental): Perifosine 209: A Phase II Trial of Perifosine in Patients with Sarcomas. Perifosine 900 mg weekly (This dose should be divided so that the maximum dose rate is 300 mg in any 4-hour interval).
  Interventions: Drug: Perifosine

INTERVENTIONS:
Drug: Perifosine — All patients should continue therapy on their current regimen until disease progression. The trial specific intervention is specified in the arms descriptions.
  Other Names: D-21266; KRX-0401
Drug: Trastuzumab — Trastuzumab was given 6mg/kg i.v. daily or 2 mg/kg i.v. on day 1, 8 and 15.
  Arms: Perifosine 206
Drug: Tamoxifen — Endocrine therapy with tamoxifen will be evaluated in combination with perifosine to determine if the combination overcomes resistance to endocrine therapy .
  Arms: Perifosine 208

SUMMARY:
This is an open label trial for patients currently enrolled in other perifosine trials.

DETAILED DESCRIPTION:
Perifosine is an oral anticancer agent with limited toxicity and a novel mechanism of action that is distinctly different from cytotoxic chemotherapies. It has been shown to inhibit and otherwise modify signaling through a number of pathways including Akt, p21, and JNK. Perifosine has been tested in Phase I and Phase II settings in a variety of dosing schedules including daily, weekly, and daily following a loading dose. In general, it has been well tolerated with dose-related nausea, vomiting, diarrhea, and fatigue being the most commonly observed toxicities.

Perifosine has induced partial responses or stable disease in solid tumors including but not limited to renal cell, sarcoma, and hepatocellular carcinoma. Perifosine is currently being studied in multiple diseases as a single agent as well as in combination with other cancer therapies. As studies are closed there are patients that have achieved a partial response or stable disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be currently receiving treatment with perifosine on a previously approved protocol.
* Patients must have had at least one evaluation following the initiation of treatment and have stable disease, partial response or complete response.
* Patient is willing to sign a new consent Regarding the protocol no exclusion criteria are described.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability | 12 weeks
  To evaluate the safety and tolerability of perifosine as a single agent as well as in combination with hormonal therapies or trastuzumab.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Grossman, MD, Study Chair — Keryx Biopharmaceuticals, Inc., NY 10022-9819